CLINICAL TRIAL: NCT03173625
Title: Single-center, Double-blind, Placebo-controlled, Randomized, Single-ascending Dose Study to Investigate the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics of AC-076 in Healthy Male Subjects
Brief Title: A Study Conducted in Healthy Male Subjects to Investigate the Safety and Tolerability of AC-76, Its Fate in the Body, and Its Effect on the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AC-076-102
Record Dates: First submitted 2017-05-23; First posted 2017-06-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AC-076 sc administration - single ascending dose (Experimental): On Day 1, 48 subjects will receive AC-076 at different single dose levels in a sequential manner and in a maximum of 6 dose levels, starting from 1 mg. Subjects will be followed by an observation period of 48 h. Each dose level will be investigated in a new group of 8 healthy male subjects (6 on active drug and 2 on placebo)
  Interventions: Drug: AC-076 for s.c. administration
- Placebo (Placebo Comparator): For each AC-076 dose level tested, 2 healthy male subjects will receive matching placebo in the same condition
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AC-076 for s.c. administration — Lyophilized AC-076A to be reconstituted with 1 mL of water for injection
  Arms: AC-076 sc administration - single ascending dose
Drug: Placebo — Sterile 0.9% w/v sodium chloride solution
  Arms: Placebo

SUMMARY:
The main objective of the study is to investigate the safety and tolerability of single ascending doses of AC-076 administered as subcutaneous injection

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Body mass index (BMI) of 18.0 to 31.0 kg/m2 (inclusive) at screening
* Systolic blood pressure (SBP) 100-145 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and pulse rate 45-90 beats per minute (inclusive) at screening
* Healthy on the basis of physical examination, electrocardiogram and laboratory tests
* Maximum (at peak) platelet aggregation ≥ 40%
* Values of closure time tested with the Platelet Function Analyzer (PFA) equipment, for both cartridges of collagen/epinephrine and collagen/ADP below the upper limit of normal range at screening

Exclusion Criteria:

* Known hypersensitivity to AC-076 or drugs of the same class, or any of their excipients
* Family or personal history of prolonged bleeding or bleeding disorders, intracranial vascular diseases, stroke, reasonable suspicion of vascular malformations, or peptic ulcers
* Platelet count < 120 × 109 L-1 at screening
* Known platelet disorders
* Orthostatic hypotension at screening (i.e., decrease from supine to standing BP of > 20 mmHg in SBP or > 10 mmHg in DBP after being in standing position for 3 min)
* Previous treatment with acetylsalicylate, non-steroidal anti-inflammatory drugs or any medication with blood thinning activity within 3 weeks prior to study drug administration; or with any other prescribed medications (including vaccines) or over the counter medications within 2 weeks prior to study drug administration
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2017-04-15 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From study treatment administration up to day 3
  Treatment-emergent AEs and treatment-emergent serious AEs
Changes from baseline in electrocardiogram (ECG) variables | From study treatment administration up to day 3
  ECG variables are to be recorded at rest using a standard 12-lead ECG
Changes from baseline in supine blood pressure | From study treatment administration up to day 3
  Supine blood pressure (mmHg)
Changes from baseline in pulse rate | From study treatment administration up to day 3
  Pulse rate (bpm)

SECONDARY OUTCOMES:
Measurement of inhibition of platelet aggregation (IPA) using anticoagulant assays | From baseline up to day 3
  Maximum (MPA) and final (FPA) platelet aggregation using light transmission aggregometry (LTA) assay.
  % inhibition of platelet aggregation (IPA), MPA and FPA.
  P2Y12 reaction units (PRU) using the VerifyNow P2Y12 assay.
  * IPA PRU
Maximum plasma concentration (Cmax) of AC-076 | From baseline up to day 3
  Cmax of AC-076 will be derived by non-compartmental analysis of the plasma concentration-time profile
time to reach Cmax (tmax) | From baseline up to day 3
  tmax of AC-076 will be derived by non-compartmental analysis of the plasma concentration-time profile
terminal half-life (t1/2) | From baseline up to day 3
  t1/2 of AC-076 will be derived by non-compartmental analysis of the plasma concentration-time profile
Area under the plasma concentration-time curves during a dosing interval [AUC(0-t)] of | From baseline up to day 3
  AUC(0-t) of AC-076 will be derived by non-compartmental analysis of the plasma concentration-time profile
Area under the plasma concentration-time curves from time 0 to inf [AUC(0-inf)] | From baseline up to day 3
  AUC(0-inf) of AC-076 will be derived by non-compartmental analysis of the plasma concentration-time profile

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- Biotrial Inc., Newark, New Jersey, United States